CLINICAL TRIAL: NCT06480240
Title: A Phase 1/2, Open-Label, Dose-Escalation and Cohort-Expansion Study Evaluating the Safety, Pharmacokinetics, and Therapeutic Activity of OBI-992 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1/2 Study of OBI-992 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-992-001
Record Dates: First submitted 2024-06-18; First posted 2024-06-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation: Interval (3+3) model
  Cohort expansion: parallel-group with randomized dosage optimization
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1 Dose Escalation - Cohort 1 (Experimental): OBI-992 at dose level 1 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 1 Dose Escalation - Cohort 2 (Experimental): OBI-992 at dose level 2 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 1 Dose Escalation - Cohort 3 (Experimental): OBI-992 at dose level 4 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 1 Dose Escalation - Cohort 4 (Experimental): OBI-992 at dose level 6 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 1 Dose Escalation - Cohort 5 (Experimental): OBI-992 at dose level 8 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 1 Dose Escalation - Cohort 6 (Experimental): OBI-992 at dose level 10 mg/kg, Q3W
  Interventions: Drug: OBI-992
- Phase 2 Cohort Expansion - Cohort 1a (Experimental): Non-small cell lung cancer indication cohort - Randomized dose optimization cohort. Dose level to be determined by the Safety Review Committee based on data available.
  Interventions: Drug: OBI-992
- Phase 2 Cohort Expansion - Cohort 1b (Experimental): Non-small cell lung cancer indication cohort - Randomized dose optimization cohort. Dose level to be determined by the Safety Review Committee based on data available.
  Interventions: Drug: OBI-992
- Phase 2 Cohort Expansion - Cohort 2 (Experimental): Small cell lung cancer indication cohort - OBI-992 dosed at putative recommended phase 2 dose.
  Interventions: Drug: OBI-992
- Phase 2 Cohort Expansion - Cohort 3 (Experimental): Gastric cancer indication cohort - OBI-992 dosed at putative recommended phase 2 dose.
  Interventions: Drug: OBI-992

INTERVENTIONS:
Drug: OBI-992 — OBI-992 is an antibody-drug conjugate

SUMMARY:
This is a 2-part trial: Part A (Dose Escalation) is designed to establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of OBI-992 (Anti-TROP2 antibody drug conjugate, anti-TROP2 monoclonal antibody-cleavable peptide linker-exatecan) as monotherapy. Part B (Cohort Expansion) is intended to further characterize the safety and preliminary clinical activity profile of the RP2D of OBI-992 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years of age or older at the time of consent
2. Provide written informed consent prior to performing any study-related procedure
3. Histologically or cytologically confirmed subjects with metastatic or advanced solid tumor that is not curable with local therapies
4. Subjects must have been treated with established standard-of-care therapy, or physicians have determined that such established therapy is not sufficiently efficacious, or subjects have declined to receive standard-of-care therapy. In the latter case, the informed consent must state the effective therapies the subject is declining.
5. Measurable disease (i.e., at least one measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1])
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ function defined as:

   a. Hepatic: i. Serum alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN), ≤5 × ULN in the presence of liver metastases ii. Serum aspartate aminotransferase (AST) ≤3 × ULN, ≤5 × ULN in presence of liver metastases iii. Serum bilirubin ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis) b. Renal: i. Creatinine clearance >50 mL/minute using Cockcroft Gault equation c. Hematologic: i. Absolute neutrophil count ≥1,500/μL ii. Platelets ≥100,000/μL iii. Hemoglobin ≥8 g/dL
8. Subjects are willing and able to comply with all protocol-required assessments, visits, and procedures, including pretreatment tumor biopsy. Archival tumor biopsies are acceptable at baseline.
9. Females of childbearing potential must have negative serum pregnancy test prior to starting study therapy and agree to use a reliable form of contraceptive during the study treatment period and for at least 120 days following the last dose of study drug. Subject not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in the trial. Postmenopausal is defined as 12 months with no menses without an alternative medical cause. Male subjects must agree to use an adequate method of contraception during the study treatment period and for at least 120 days following the last dose of study drug.
10. Cannot be breast feeding
11. Subjects with human immunodeficiency virus (HIV) infection are eligible if CD4+ Tcell counts ≥ 350 cells/μL; subjects on anti-retroviral therapy (ART) should be on an established dose for at least 4 weeks and have an HIV viral load less than 200 copies/mL prior to enrollment.
12. Subjects with serological evidence of chronic hepatitis B virus (HBV) infection are eligible if they have an HBV viral load below the limit of quantification with or without concurrent viral suppressive therapy.
13. Subjects with a history of hepatitis C virus (HCV) infection can be under curative antiviral treatment and have a viral load below the limit of quantification.
14. Subjects in Part B (Cohort-Expansion) - must have one of the following tumor types to be enrolled in the respective cohort:

    * Cohort 1: Non-small cell lung cancer (NSCLC)

      o Pathologically confirmed subjects with metastatic NSCLC with or without actionable genomic alterations.
    * Cohort 2: Small cell lung cancer (SCLC)
    * Cohort 3: Gastric cancer

Exclusion Criteria:

1. Less than 3 weeks from prior cytotoxic chemotherapy or radiation therapy; and less than 5 half-lives or 3 weeks, whichever is shorter, from prior biologic therapies, prior to the first dose of OBI-992
2. Has undergone a major surgical procedure (as defined by the Investigator) or significant traumatic injury within 28 days prior to the first dose of OBI-992
3. Sensory or motor neuropathy of Grade 2 or greater
4. Subjects with a history of solid organ transplant
5. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), except for alopecia and laboratory values listed in the inclusion criteria
6. Corrected QT interval (QTcF) prolongation to >470 msec based on the average of the screening 12-lead ECGs
7. Known hypersensitivity to OBI-992 or its excipients
8. Has known untreated central nervous system (CNS) metastases. Subjects with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period
9. Has significant clinical cardiac abnormality (e.g., clinical heart failure or unstable angina)
10. Any medical comorbidity that is life-threatening or, in the opinion of the Investigator, renders the subject unsuitable for participation in a clinical trial due to possible noncompliance, would place the subject at an unacceptable risk (e.g. Interstitial lung disease (ILD)) and/or potential to affect interpretation of results of the study.
11. Subjects in Part B (Phase 2 Cohort Expansion) may not have had prior therapy with an approved or investigational TROP2 ADC (prior TROP2 ADC therapy allowed during dose escalation)
12. Is receiving any concurrent prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of OBI-992: incidence of adverse events, serious adverse events, and laboratory abnormalities | Duration of study, up to 2 years and 2 months
  To determine the safety and tolerability of OBI-992 when administered to subjects with advanced solid tumors, based on adverse events (AEs), serious adverse events (SAEs) and laboratory abnormalities graded by NCI CTCAE v5.0
Maximum tolerated dose and recommended Phase 2 dose of OBI-992 | Duration of study, up to 2 years and 2 months
  To determine the maximum tolerated dose (MTD) and optimal recommended phase 2 dose (RP2D) of OBI-992
Preliminary clinical activity profile - objective response rate (ORR) | Duration of study, up to 2 years and 2 months
  Percentage of subjects in the as-treated population with objective response according to response evaluation criteria in solid tumors (RECIST v.1.1)
Preliminary clinical activity profile - clinical benefit rate (CBR) | Duration of study, up to 2 years and 2 months
  Percentage of subjects in the as-treated population with clinical benefit according to response evaluation criteria in solid tumors (RECIST v.1.1)
Preliminary clinical activity profile - duration of response (DOR) | Duration of study, up to 2 years and 2 months
  Percentage of subjects in the as-treated population with response according to response evaluation criteria in solid tumors (RECIST v.1.1)
Preliminary clinical activity profile - disease control rate (DCR) | Duration of study, up to 2 years and 2 months
  Percentage of subjects in the as-treated population with disease control according to response evaluation criteria in solid tumors (RECIST v.1.1)
Preliminary clinical activity profile - progression-free survival | Duration of study, up to 2 years and 2 months
  Percentage of subjects in the as-treated population with progression-free survival according to response evaluation criteria in solid tumors (RECIST v.1.1)

SECONDARY OUTCOMES:
Immunogenicity of OBI-992: anti-drug antibodies (ADAs) | Duration of study, up to 2 years and 2 months
  To evaluate the immunogenicity of OBI-992 (anti-drug antibodies), characterized by percentage of subjects with ADAs in blood
Serum pharmacokinetics (PK): Peak Plasma Concentration (Cmax) of OBI-992 and its active metabolite | Duration of study, up to 2 years and 2 months
  To determine the serum Cmax of OBI-992 and its active metabolite exatecan
Serum pharmacokinetics (PK): area under the concentration-time curve (AUC) of OBI-992 and its active metabolite | Duration of study, up to 2 years and 2 months
  To determine the serum AUC of OBI-992 and its active metabolite exatecan
Serum pharmacokinetics (PK): half-life (T1/2) of OBI-992 and its active metabolite | Duration of study, up to 2 years and 2 months
  To determine the serum half-life of OBI-992 and its active metabolite exatecan
Serum pharmacokinetics (PK): clearance (CL) of OBI-992 and its active metabolite | Duration of study, up to 2 years and 2 months
  To determine the serum clearance (CL) of OBI-992 and its active metabolite exatecan
Serum pharmacokinetics (PK): Volume distribution at steady state (Vdss) of OBI-992 and its active metabolite | Duration of study, up to 2 years and 2 months
  To determine the serum volume distribution at steady state of OBI-992 and its active metabolite exatecan

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - California Clinical Trials Medical Group (CCTMG), Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- Taiwan (2):
  - Taipei Tzu Chi Hospital, New Taipei City, Xindian District
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City, Zhonghe District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shia CS, Wen SN, Hsu RY, Tu JS, Chang HW, Weng HC, Yang JJ, Chiang MF, Tsao YH, Lu CH, Chen YH, Wu YC, Chen YC, Li WF, Huang TY, Lai MT. Preclinical Pharmacokinetic, Pharmacodynamic, and Safety Profile of OBI-992: A Novel TROP2-Targeted Antibody-Drug Conjugate. Mol Cancer Ther. 2025 Dec 2;24(12):1938-1947. doi: 10.1158/1535-7163.MCT-24-1176. PMID 40762235